CLINICAL TRIAL: NCT05986916
Title: Accurate Point of Care Liver Disease Diagnostics
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Livivos, Inc. (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Claude Sirlin, Professor of Radiology, University of California, San Diego
Other Study IDs: 806222; 1R43DK135225-01 (NIH); 1R43EB034626-01A1 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: NAFLD; Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection; Body Weights and Measures; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single arm: This is a single arm study in which all participants undergo the same research procedures.
  Interventions: Diagnostic Test: Liverscope® exam; Diagnostic Test: MR exam; Diagnostic Test: FibroScan® exam (optional); Other: Blood draw; Other: Body measurements; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Liverscope® exam — Participants will undergo a LiverScope® examination to measure liver proton density fat fraction (PDFF, primary) and T1 and T2 values (exploratory).
Diagnostic Test: MR exam — Participants will undergo an advanced MR examination to measure liver PDFF, T1, T2, and liver stiffness values.
Diagnostic Test: FibroScan® exam (optional) — Participants may undergo a FibroScan® exam (optional) to evaluate liver fat and liver stiffness.
Other: Blood draw — Participants will undergo a blood draw (approximately 10 mL) for measurement of CBC, platelets, and complete metabolic panel with transaminases.
Other: Body measurements — Participants will have their height, weight, waist circumference, and hip circumference measured.
Other: Questionnaires — Participants will be asked to fill out questionnaires to collect information about their alcohol consumption, history of cigarette smoking, presence of diabetes, and history of liver disease and medications

SUMMARY:
This research study is being conducted to find out more about techniques to non-invasively evaluate liver disease. The investigators are testing a new technology to evaluate the liver (LiverScope®), and they will compare it to other methods to evaluate the liver, including advanced conventional liver MR and liver FibroScan® ultrasound exams. MR exams and FibroScan® ultrasound exams are common exams used to monitor NAFLD. Conventional MR scanners use magnetic fields and radio waves to make pictures of the liver. LiverScope® is a small, portable MR-based device that uses similar, but simplified technology, and can be used on top of an exam table in an outpatient setting. LiverScope® currently is not approved for clinical use.

In this study the investigators will learn how LiverScope® measurements of the liver compare to MR.

Study participants will be asked to complete a one-time visit which includes:

* LiverScope exam
* MR exam
* FibroScan exam (optional)
* Blood draw
* Completion of study questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age:18 years or older
* Known or clinically suspected NAFLD
* Weight less than 350 lbs (safety limit of MR scanner table)
* Able to lie on LiverScope® diagnostic table for about 15 min
* Able to hold breath repeatedly for about 20 s during MR and LiverScope® exams
* Willing and able to undergo all study procedures

Exclusion Criteria:

* VA patient only; not a UCSD patient
* UCSD or Livivos study personnel
* MR contraindication(s)
* Potential participant states that she knows that she is pregnant, thinks she may be pregnant or states she is trying to become pregnant*
* Known chronic liver disease other than NAFLD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinically known or suspected liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Repeatability and reproducibility coefficients of LiverScope® PDFF measurements | Up to 3 months
  Estimation of repeatability and reproducibility coefficients of liver PDFF values measured by LiverScope®.
Agreement of LiverScope® PDFF measurements with MRI PDFF measurements | Up to 3 months
  Assessment of the agreement between LiverScope® PDFF measurements and MRI PDFF measurements.

SECONDARY OUTCOMES:
Repeatability and reproducibility coefficients of LiverScope® T1 measurements | Up to 3 months
  Estimation of repeatability and reproducibility coefficients of liver T1 values estimated by LiverScope®.
Correlation coefficient between LiverScope® T1 and T2 measurements and MRS T1 and T2 measurements | Up to 3 months
  Estimation of the correlation coefficient between LiverScope® T1 and T2 measurements and MRS T1 and T2 measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Claude B Sirlin, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This is an SBIR study. De-identified coded data will be shared as per grant application.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after completion
Access Criteria: Public
URL: https://library.ucsd.edu/dc